CLINICAL TRIAL: NCT05507398
Title: Comparative Clinical Study Evaluating the Anti-tumor Effect of Metformin Versus Atorvastatin as an Adjuvant Therapy With Chemotherapy in Patients With Non-metastatic Breast Cancer
Brief Title: The Anti-tumor Effect of Metformin And Atorvastatin in Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Mohammed El-Abd, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breast cancer treatment
Record Dates: First submitted 2022-08-14; First posted 2022-08-19 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Metformin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): 30 patients who will serve as a control group and will receive placebo tablets
  Interventions: Drug: Placebo, metformin and atorvastatin
- metformin group (Active Comparator): 30 patients who will receive metformin 1000 mg/day.
  Interventions: Drug: Placebo, metformin and atorvastatin
- atorvastatin group (Active Comparator): 30 patients who will receive atorvastatin 20 mg/day.
  Interventions: Drug: Placebo, metformin and atorvastatin

INTERVENTIONS:
Drug: Placebo, metformin and atorvastatin — comparing the anti-tumor effects of metformin and atorvastatin
  Other Names: Cidophage 1000 mg; Ator 20 mg

SUMMARY:
This study aims at evaluating and comparing the anti-tumor effects of metformin and statins (hydroxyl-methyl-glutaryl-CoA reductase inhibitors) in patients with non-metastatic breast cancer (stage I, II, & III).

DETAILED DESCRIPTION:
Worldwide, BC is the most frequently diagnosed life-threatening cancer in women. In EGYPT, breast cancer is the foremost oncologic problem, contributing to 20% of all cancers and 43% of female cancers. Metformin and atorvastatin have anti-tumor effects. To date, there are limited data to investigate and compare the anti-tumor effect between metformin and statins in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologically and histologically (biopsy) confirmed diagnosis of breast cancer and with stage I, II, and stage III breast cancer according to the American Joint Committee on Cancer (TNM staging system of breast cancer).
* Patients with no contraindication for chemotherapy, metformin, or statins
* Females aged ≥ 18 years old
* Performance status < 2 according to the Eastern Cooperative Oncology Group (ECOG) score

Exclusion Criteria:

* Patients with metastatic breast cancer (stage IV)
* Pregnant or lactating women.
* Patients with hepatic or renal impairment.
* Patients with myopathy.
* Patients with any condition predispose to acidosis (COPD, heart failure, ….)
* Patients who had dementia, mental retarded, and any psychiatric condition that would prohibit the understanding or signing of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in the overall response rate | 6 months
  The improvement in the overall response rate (ORR) will be assessed in 3 arms at the end of the study using the RECIST criteria and Miller-Payne grading system respectively
Improvement in the pathological response | 6 monthes
  The improvement in the pathological response will be assessed in 3 arms at the end of the study using the RECIST criteria and Miller-Payne grading system respectively

CONTACTS AND LOCATIONS:
Overall Officials: ahmed elabd, doctor, Principal Investigator — Tanta university, faculty of pharmacy